CLINICAL TRIAL: NCT01554397
Title: Phase II/III Clinical Trial of Intensity Modulated Radiation Therapy With Concurrent Cisplatin for Stage I-IVA Cervical Carcinoma
Brief Title: Study With Intensity Modulated Radiation Therapy With Cisplatin to Treat Stage I-IVA Cervical Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Loren Mell, MD, Associate Professor, Director Division of Clinical and Translational Research, Department of Radiation Medicine and Applied Sciences., University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INTERTECC; R21CA162718-01 (NIH)
Record Dates: First submitted 2012-03-08; First posted 2012-03-15 (Estimated); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Cervical Cancer
Keywords: Cervical; Carcinoma; Cisplatin; IMRT; Radiation; INTERTECC; International; External Beam; Brachytherapy; LDR; HDR; IGRT; CBCT
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma | interventions — Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Phase II: IMRT (standard) vs. PET-guided Bone Marrow-Sparing IMRT (experimental), non-randomized Phase III: IMRT (standard) vs. PET-guided Bone Marrow-Sparing IMRT (experimental), randomized
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMRT with concurrent cisplatin 40 mg/m2 (Active Comparator): Intensity-modulated Radiation Therapy (IMRT) with concurrent cisplatin 40 mg/m2
  Interventions: Drug: Cisplatin; Radiation: IMRT
- PET-guided Bone Marrow-Sparing IMRT (Experimental): PET-guided Bone Marrow-Sparing IMRT with concurrent cisplatin 40 mg/m2
  Interventions: Radiation: PET-guided Bone Marrow-Sparing Intensity Modulated Radiation Therapy (IMRT); Drug: Cisplatin

INTERVENTIONS:
Radiation: PET-guided Bone Marrow-Sparing Intensity Modulated Radiation Therapy (IMRT) — IMRT 45.0 Gy (intact) or 50.4 Gy (postoperative high-risk) in 1.8 Gy daily fractions over 5-5.5 weeks with PET-guided Bone Marrow-Sparing
  Other Names: PET-guided Bone Marrow-Sparing IMRT
  Arms: PET-guided Bone Marrow-Sparing IMRT
Drug: Cisplatin — Weekly infusion of 40 mg/m2 (80 mg max) x 5 weeks
  Other Names: Platinol
Radiation: IMRT — IMRT 45.0 Gy (intact) or 50.4 Gy (postoperative high-risk) in 1.8 Gy daily fractions over 5-5.5 weeks
  Other Names: Intensity Modulated Radiation Therapy
  Arms: IMRT with concurrent cisplatin 40 mg/m2

SUMMARY:
The purpose of this study is to find out whether patients with cervical cancer treated with PET-guided Bone Marrow Sparing IMRT have less side effects with equal cancer control compared to standard radiation techniques (IMRT). The hypothesis is that PET-guided Bone Marrow Sparing IMRT will reduce acute hematologic and gastrointestinal toxicity and increase chemotherapy tolerance for cervical cancer patients treated with concurrent cisplatin.

DETAILED DESCRIPTION:
Multiple randomized controlled trials have established concurrent cisplatin-based chemoradiotherapy as the standard of care for locally advanced cervical cancer [3-8]. The addition of concurrent cisplatin to radiotherapy (RT) increases pelvic control, disease-free survival (DFS) and overall survival; however, 5-year DFS and overall survival are still only approximately 60% and 5-year pelvic failure is approximately 30%. Moreover, acute gastrointestinal (GI) and hematologic toxicity are increased. Approximately 30% of patients will experience acute grade ≥ 3 toxicity, predominantly GI and hematologic. Methods to reduce toxicity during chemoradiotherapy, particularly gastrointestinal and hematologic, could mitigate this toxicity and take advantage of the therapeutic benefits of intensive concurrent chemotherapy.

Intensity modulated radiation therapy (IMRT) is a modern RT technique that differs from conventional techniques in many ways. First, patients undergo computed tomography (CT) simulation so that customized target volumes can be defined 3-dimensionally. IMRT treatment planning involves multiple beam angles and uses computerized inverse treatment planning optimization algorithms to identify dose distributions and intensity patterns that conform dose to the target, reducing radiation dose to surrounding tissues. IMRT delivery is typically accomplished with the use of multileaf collimators, which involve small motorized leaflets (collimators) that move in and out of the beam path, modulating the dose intensity.

PET-guided Bone Marrow Sparing IMRT is designed to spare hematopoietically active subregions of the pelvic bone marrow using quantitative image segmentation. Previous studies indicate this approach can reduce toxicity and improve chemotherapy tolerance, which may improve outcomes and help optimized delivery of cytotoxic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven, invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix
* Biopsy result positive for carcinoma within 60 days prior to registration
* FIGO clinical stage I-IVA disease, based on standard diagnostic workup, including:History/physical examination and/or Examination under anesthesia (if indicated)
* If the patient is status post hysterectomy, one or more of the following conditions must be present: positive lymph nodes, positive margins, parametrial invasion, or non-radical surgery (i.e., simple hysterectomy).
* If the patient is inoperable, one or more of the following conditions must be present: clinical stage IB2-IVA, positive lymph nodes on nodal sampling or frozen section, and/or parametrial invasion
* Within 42 days prior to registration, the patient must have any of the following, if clinically indicated: examination under anesthesia, cystoscopy, sigmoidoscopy, rigid proctoscopy, or colonoscopy.
* X-ray (PA and lateral), CT scan, or PET/CT scan of the chest within 42 days prior to registration;
* CT scan, MRI, or PET/CT of the pelvis within 42 days prior to registration;
* Karnofsky Performance Status 60-100
* Absolute neutrophil count (ANC) ≥ 1500 cells/mm3; Platelets ≥ 100,000 cells/mm3; Hemoglobin ≥ 10.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10.0 g/dl is acceptable); Creatinine clearance ≥ 50 mg/dl; Bilirubin < 1.5 mg/dl; WBC ≥ 3,000/μl; ALT/AST < 3 x ULN; INR ≤ 1.5
* Negative serum pregnancy test for women of child-bearing potential

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer), unless disease free for a minimum of 3 years;
* Prior systemic chemotherapy within the past three years
* Prior radiotherapy to the pelvis or abdomen that would result in overlap of radiation therapy fields;
* Para-aortic, inguinal, or gross (unresected) pelvic nodal metastasis. Gross pelvic nodal metastasis is defined as either: Radiographic evidence of nodal metastasis on CT or MRI (node having short axis diameter > 1 cm)OR Radiographic evidence of nodal metastasis on diagnostic FDG-PET or PET/CT scan (abnormally increased FDG uptake as determined and documented by the radiologist)OR Biopsy-proven metastasis (e.g. needle biopsy) in undissected node
* Distant metastasis
* Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* Uncontrolled diabetes, defined as diabetes mellitus, which in the opinion of any of the patient's physicians requires an immediate change in management;
* Uncompensated heart disease or uncontrolled high blood pressure
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-10-13 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loren Mell, MD, Principal Investigator — University of California, San Diego
Locations (7):
- United States (2):
  - Moores UC San Diego Cancer Center, La Jolla, California
  - University of Miami Miller School of Medicine, Miami, Florida
- Xijing Hospital, Xi'an, China
- University Hospital Hradec Králové, Hradec Králové, Czechia
- Tata Memorial Hospital, Pārel, Mumbai, India
- Marie Sklodowska Cancer Center, Gliwice, Poland
- King Chulalongkorn Hospital, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 participants determined to be ineligible. 1 participant withdrew before protocol therapy due to an emergency
Groups:
- IMRT: IMRT with concurrent cisplatin 40 mg/m2
  Intensity Modulated Radiation Therapy (IMRT): 45.0 Gy (intact) or 50.4 Gy (postoperative high-risk) in 1.8 Gy daily fractions over 5-5.5 weeks
  Cisplatin: Weekly infusion of 40 mg/m2 (80 mg max) x 5 weeks
- PET-Guided Bone Marrow-Sparing IMRT: PET-Guided Bone Marrow-Sparing IMRT with concurrent cisplatin 40 mg/m2
  Intensity Modulated Radiation Therapy (IMRT): 45.0 Gy (intact) or 50.4 Gy (postoperative high-risk) in 1.8 Gy daily fractions over 5-5.5 weeks
  Cisplatin: Weekly infusion of 40 mg/m2 (80 mg max) x 5 weeks
Period: Overall Study
Arm/Group | IMRT | PET-Guided Bone Marrow-Sparing IMRT
Started | 63 | 46
Completed | 55 | 46
Not Completed | 8 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ineligible | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- IMRT: All patients receive IMRT with concurrent cisplatin 40 mg/m2
  Intensity Modulated Radiation Therapy (IMRT): 45.0 Gy (intact) or 50.4 Gy (postoperative high-risk) in 1.8 Gy daily fractions over 5-5.5 weeks
  Cisplatin: Weekly infusion of 40 mg/m2 (80 mg max) x 5 weeks
- Total: Total of all reporting groups
Arm/Group | IMRT | PET-Guided Bone Marrow-Sparing IMRT | Total
Number analyzed (Participants) | 55 | 46 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (12.9) | 46 (51.2) | 52.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 46 | 101
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 49 | 33 | 82
  Unknown or Not Reported | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 0 | 0 | 0
  Asian | 11 | 7 | 18
  Latina/Hispanic | 3 | 9 | 12
  White, non-Hispanic | 38 | 26 | 64
  Other/unknown | 3 | 4 | 7
Kamofsky Status [Count of Participants; unit: Participants] — The Karnofsky status will be used to measure quality of life and the ability to carry out every day tasks. The higher the score, the more the patient is able to do based on the below scale:
  100-Normal no complaints; no evidence of disease 90-Able to carry on normal activity; minor signs or symptoms of disease 80-Normal activity with effort; some signs or symptoms of disease
  Participants
    70 | 0 | 1 | 1
    80 | 4 | 1 | 5
    90 | 22 | 17 | 39
    100 | 29 | 27 | 56
Grade [Count of Participants; unit: Participants] — Grade describes how differentiated cells are from typical cells. The more the cancer cells look like typical cells, the lower the grade.
  * grade 1 (low grade)- some abnormalities but similar looking to a typical cell
  * grade 2 (moderate grade)- moderate abnormalities
  * grade 3 (high grade) highly abnormal and do not look like typical cells
  Participants
    1 | 3 | 1 | 4
    2 | 28 | 16 | 44
    3 | 18 | 16 | 34
    Not graded | 6 | 13 | 19
Figo Stage [Count of Participants; unit: Participants] — Doctors assign the FIGO stage of the cancer by evaluating the tumor and whether the cancer has spread to other parts of the body.
  FIGO staging is based on a the results of a physical exam, imaging scans, and biopsies. Stage I-IV with Stage I being confined to the cervix and Stage IV resulting in spread to adjacent or distant organs.
  Participants
    IB1 | 1 | 3 | 4
    IB2 | 5 | 7 | 12
    IIA1 | 3 | 1 | 4
    IIB | 41 | 25 | 66
    IIIB | 3 | 10 | 13
    IVA | 2 | 0 | 2
Histologic Status [Count of Participants; unit: Participants]
  Squamous cell Carcinoma | 47 | 36 | 83
  Adenocarcinoma | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Primary Event (Acute Hematologic or GI Toxicity)
Description: Acute grade >= 3 neutropenia or clinically significant >=2 diarrhea or any grade >=3 GI toxicity
Time Frame: Up to 30 days post radiation, about one month
Measure: Count of Participants; unit: Participants
Groups:
- IMRT Arm (Phase II): IMRT with concurrent cisplatin 40 mg/m2
  Cisplatin: Weekly infusion of 40 mg/m2 (80 mg max) x 5 weeks
- PET-Guided BMS-IMRT (Phase II): PET-Guided BMS-IMRT with concurrent cisplatin 40 mg/m2
  Intensity Modulated Radiation Therapy (IMRT): 45.0 Gy (intact) or 50.4 Gy (postoperative high-risk) in 1.8 Gy daily fractions over 5-5.5 weeks
  Cisplatin: Weekly infusion of 40 mg/m2 (80 mg max) x 5 weeks
Arm/Group | IMRT Arm (Phase II) | PET-Guided BMS-IMRT (Phase II)
Number analyzed (Participants) | 55 | 46
Participants | 55 | 46

2. Secondary Outcome: Progression-free Survival
Description: Time from registration to first recurrence of disease or death from any cause
Time Frame: Up to 36 Months post treatment, a total of about 38 months
Measure: Count of Participants; unit: Participants
Groups:
- PET-Guided Bone Marrow-Sparing IMRT: All patients receive PET-Guided Bone Marrow-Sparing IMRT with concurrent cisplatin 40 mg/m2
  Intensity Modulated Radiation Therapy (IMRT): 45.0 Gy (intact) or 50.4 Gy (postoperative high-risk) in 1.8 Gy daily fractions over 5-5.5 weeks
  Cisplatin: Weekly infusion of 40 mg/m2 (80 mg max) x 5 weeks
Arm/Group | PET-Guided Bone Marrow-Sparing IMRT | IMRT
Number analyzed (Participants) | 46 | 55
Participants | 46 | 55

3. Secondary Outcome: Acute Adverse Events
Description: Acute grade 2 and 3 Adverse Events occurring Up to 30 days post-treatment
Time Frame: Up to 30 days post-treatment, about one month
Measure: Number; unit: participants
Arm/Group | PET-Guided Bone Marrow-Sparing IMRT | IMRT
Number analyzed (Participants) | 46 | 55
participants
  Grade 2 or higher GI toxicity | 17 | 17
  Grade 3 or higher GI toxicity | 2 | 1
  Grade 3 or higher hematologic toxicity | 17 | 25

ADVERSE EVENTS:
Time Frame: 38 months
Arm/Group | IMRT | PET-Guided Bone Marrow-Sparing IMRT
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/46
Other Adverse Events (participants affected / at risk) | 55/55 | 46/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMRT (N=55) | PET-Guided Bone Marrow-Sparing IMRT (N=46)
Clinically significant GI toxicity (Gastrointestinal disorders) | 18 (18) | 19 (19)
Grade 3 or higher neutropenia (Investigations) | 50 (50) | 28 (28)
Grade 2 GI toxicity (Gastrointestinal disorders) | 17 (17) | 17 (17)
Grade 3 or higher GI toxicity (Gastrointestinal disorders) | 1 (1) | 2 (2)
Grade 3 or higher hematologic toxicity (Investigations) | 25 (25) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT01554397/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT01554397/ICF_001.pdf